CLINICAL TRIAL: NCT04481516
Title: Effect of Breathing-based Meditation (Sudarshan Kriya Yoga) in NHS Health Care Workers With Possible COVID-19 Related Stress and Anxiety Disorder
Brief Title: Yoga in NHS Health Care Workers With COVID-19 Related Stress
Status: Withdrawn | Type: Observational
Why Stopped: Put on hold due to COVID and then withdrawn.
Sponsor: Doncaster And Bassetlaw Hospitals NHS Foundation Trust (Other)
Responsible Party: Sponsor
Other Study IDs: DBH 1058/2020/HRAS
Record Dates: First submitted 2020-07-01; First posted 2020-07-22 (Actual); Last update posted 2024-07-08 (Actual); Status verified 2021-06

CONDITIONS: Stress
Keywords: Stress; Yoga
MeSH Terms: interventions — Yoga

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Yoga: Single group study representing cohort of NHS health care workers with possible Covid-19 related stress and anxiety disorder. Participants act as their own controls pre and post regular practice of yoga technique.
  Interventions: Other: Yoga

INTERVENTIONS:
Other: Yoga — SKY Yoga

SUMMARY:
Recent reports have highlighted Covid-19 related increase in levels of depression and stress related disorders in the health care professionals. Pranayama (ancient yogic breathing techniques) helps harmonizing breathing by regular voluntary control of breath.

Yoga has been shown to modulate autonomic nervous functions of the brain. Sudarshan kriya Yoga (SKY) is a unique form of pranayama taught by ''Art of Living UK'' a non-profit organization -for over two decades. SKY involves simple rhythmic breathing technique (easy to practice) that aims at harmonizing body, mind and emotions. Sudarshan kriya yoga (SKY) has been shown to be beneficial in reducing levels of stress, anxiety and depression. This breathing based meditation technique has previously been shown to be beneficial in post-traumatic stress disorder.

In this pilot study the aim is to assess the feasibility and effect of SKY in NHS health care workers with possible Covid-19 related stress and anxiety disorder.

DETAILED DESCRIPTION:
In the current pilot study the aim is to assess the feasibility and effect of SKY in NHS health care workers with possible Covid related stress and anxiety disorder. Study participants are staff members of Doncaster and Bassetlaw Hospitals NHS Foundation Trust who may be affected Covid related stress and anxiety disorder.

This is a paperless study with all the information including participant information, consent forms and link to questionnaires sent via the trust e-mail.

Information about the study would be advertised via trust intranet, trust facebook page, and through flyers across various sites within the trust. Potential participants who are interested to know more information would be encouraged to contact the research team on dbth.sky.yoga@nhs.net by using their trust email.

They would then be sent a generalised anxiety disorder (GAD-7) questionnaire to answer via e-mail and they would be eligible to participate if their GAD-7 score is ≥5 which implies they have mild or more sever form of anxiety disorder.

They would then be sent an invitation letter, participant information leaflet and consent form via e-mail. They would also be provided an opportunity to talk to a research team member via telephone. They would be enrolled into the study after receipt of their consent via e-mail and they will be provided with a unique identifier number (which would be used for the rest of the study). Participants receive online tutorial on breathing based meditation (SKY) for about 4-5 hours spread over 3 sessions using Zoom platform from an 'Art of Living' certified yoga teacher. They are subsequently encouraged to practice this technique for about 20 mins a day. They are also offered an optional online group session lasting 20mins, 4 days a week for the first 6 weeks and subsequently once a week for the duration of the study.

They are sent a link, to their trust email, to access questionnaire about their symptoms and health which they will need to answer at onset, 6 weeks, 3 months and at conclusion of the study (6 months). They will need to provide personal information about their medical condition and their medications at the time of enrolment. On completion of the study results would be analysed and final outcome presented. Study findings would be disseminated in medical fraternity by presentation in medical conference and publication in a peer reviewed journal.

ELIGIBILITY:
Inclusion Criteria:

* Male / Female aged over 18 years
* Member of DBHFT
* Score of ≥ 5 on generalized anxiety disorder (GAD-7) questionnaire
* Fully able to understand the nature of the study with sufficient chance to read PIL and commitment to participate in the online Yoga schedule
* Willingness to enter data regularly by answering online questionnaire

Exclusion Criteria:

* Under 18 years of age
* Significant other co-morbid conditions that would preclude regular Yoga practice
* Chronic medical conditions necessitating hospital admission in the last 6 months or history of significant bipolar disorder
* Patients taking part in other research studies during the study period
* Inability to understand study requirements
* Patients who have been on any form of regular Yoga schedule in the previous 6 months

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: NHS staff members with self-reported stress due to COVID
Sampling Method: Non-Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2020-07-01 (Actual); Primary Completion 2021-02-28 (Actual); Study Completion 2021-12-28 (Actual)

PRIMARY OUTCOMES:
Alleviated stress 1 - short term | 6 weeks
  (1) To assess feasibility and efficacy of regularly supervised SKY in the NHS health care workers with possible Covid-19 related stress and anxiety disorder in the short term (6 weeks) by using Generalised Anxiety Disorder questionnaire score ranging from 0-21, higher score associated with worse outcome
Alleviated stress 2 - short term | 6 weeks
  (2) To assess feasibility and efficacy of regularly supervised SKY in the NHS health care workers with possible Covid-19 related stress and anxiety disorder in the short term (6 weeks) by using Medical Outcomes Study Questionnaire Short Form 36 Health Survey questionnaire score ranging from 36-149, higher score associated with worse outcome
Alleviated stress 3 - short term | 6 weeks
  (3) To assess feasibility and efficacy of regularly supervised SKY in the NHS health care workers with possible Covid-19 related stress and anxiety disorder in the short term (6 weeks) by using Patient Health Questionnaire questionnaire score ranging from 0-27, higher score associated with worse outcome

SECONDARY OUTCOMES:
Alleviated stress 1 - medium term | 3-6 months
  (1) To assess feasibility and efficacy of regularly supervised SKY in the NHS health care workers with possible Covid-19 related stress and anxiety disorder in the short term (6 weeks) by using Generalised Anxiety Disorder questionnaire score ranging from 0-21, higher score associated with worse outcome
Alleviated stress 2 - medium term | 3-6 months
  (2) To assess feasibility and efficacy of regularly supervised SKY in the NHS health care workers with possible Covid-19 related stress and anxiety disorder in the short term (6 weeks) by using Medical Outcomes Study Questionnaire Short Form 36 Health Survey questionnaire score ranging from 36-149, higher score associated with worse outcome
Alleviated stress 3 - medium term | 3-6 months
  (3) To assess feasibility and efficacy of regularly supervised SKY in the NHS health care workers with possible Covid-19 related stress and anxiety disorder in the short term (6 weeks) by using Patient Health Questionnaire questionnaire score ranging from 0-27, higher score associated with worse outcome

CONTACTS AND LOCATIONS:
Overall Officials: Venkata D Nagarajan, Principal Investigator — Doncaster and Bassetlaw Teaching Hospitals NHS Foundation Trust
Locations (1):
- Doncaster and Bassetlaw Teaching Hospitals NHS Foundation Trust, Doncaster, South Yorkshire, United Kingdom

IPD SHARING:
Plan to Share IPD: No
All data will be pseudonymised